CLINICAL TRIAL: NCT02240537
Title: Phase I Study of an Oncofetal Antigen ("OFA") Multi-Peptide Immunotherapy ("BBMPI03") in Subjects With Hematologic Cancer
Brief Title: Phase I Study of an Oncofetal Antigen Multi-Peptide Immunotherapy in Subjects With Hematologic Cancer
Acronym: BBMPI03
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Benovus Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBMPI03-Hem-01
Record Dates: First submitted 2014-09-09; First posted 2014-09-15 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Acute Myelogenous Leukemia (AML); Multiple Myeloma (MM); Myelodysplastic Syndrome (MDS); Smoldering Multiple Myeloma (sMM)
Keywords: AML; MM; MDS; sMM
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Multiple Myeloma; Myelodysplastic Syndromes; Smoldering Multiple Myeloma | interventions — sargramostim; Monatide (IMS 3015); Emulsions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label Treatment Arm (Experimental): BB-MPI-03 peptides plus montanide plus sargramostim
  Interventions: Drug: Sargramostim; Drug: BB-MPI-03; Drug: Montanide

INTERVENTIONS:
Drug: Sargramostim — Drug: Sargramostim (GM-CSF) Other Names: Leukine Sargramostim (250 ug vial) is reconstituted with 0.5 ml of Sterile Water for Injection. Subjects will receive 0.5 ml intradermally (250 µg) near the arm pit or inside of thigh.
  Other Names: Leukine
Drug: BB-MPI-03 — Other Names: Multi-peptide immunotherapy (MPI) is comprised of 3 cytotoxic T-cell epitopes derived from oncofetal antigen. There are 3 dose levels of study vaccine planned to be tested, starting at 0.25 mg each peptide (0.75 mg total peptide dose), then 0.5 mg of each peptide (1.5 mg total) and finally 1 mg each peptide (3 mg total). At the starting dose of 0.75 mg, the BB MPI 03-15 mg vial is used and 100 ul is administered; at the 1.5 mg dose, 200 ul of the BB MPI 03-15 mg vial is used; at the 3 mg dose, 200 ul of the BB MPI 03-30 mg is used.
  Other Names: Multi-peptide Immunotherapy
Drug: Montanide — Drug: Montanide Other Names: mineral oil, USP BB-MPI-03 is emulsified with Montanide and administered intradermally (ID) within 1-2 cm of the 2 sargramostim injection sites 1-3 minutes after sargramostim administration.
  Subjects and the injection sites are to be monitored for 1 hour after sargramostim and BB-MPI-03 emulsion administration.
  Other Names: Emulsion

SUMMARY:
The study is designed to evaluate safety, immunogenicity, and preliminary anti-tumor activity of a multi-peptide immunotherapy (BB-MPI-03) at three peptide+adjuvant dose levels. The peptides stimulate cytotoxic T-cells targeting oncofetal antigen (OFA). Subjects with AML, MM, sMM, or MDS who are off treatment and with stable disease or better, or who are not eligible for or refuse allogeneic HSCT are to be enrolled. The study will be conducted at 2 to 4 study centers in the US.

DETAILED DESCRIPTION:
The current study is a Phase I, open-label, multi-center, dose escalation study designed to evaluate safety, immunogencity, and potential anti-tumor activity of BB-MPI-03 at three peptide plus adjuvant dose levels. Subjects with acute myelogenous leukemia (AML), multiple myeloma (MM), smoldering multiple myeloma (sMM), or myelodysplastic syndrome (MDS) who are off treatment and with stable disease or better or who are not eligible for or refuse allogeneic hematopoietic stem cell transplantation (HSCT) are to be enrolled. The study will be conducted at 2 to 4 study centers in the United States (US).

The study employs a sequential group, open-label, 3+3 dose- escalation design to determine the safety and MTD of BB- MPI-03.

ELIGIBILITY:
Inclusion Criteria

a. History of morphologically confirmed AML w/ classification other than WHO Acute Promyelocytic Leukemia (FAB M3), based on bone marrow examination.

i. not a candidate for allogeneic HSCT or no intention to move to HSCT at time of enrollment.

ii. Patient's AML could be in morphologic CR or no further cytotoxic chemotherapy is currently being considered.

iii. Completed consolidation chemotherapy, if available and/or appropriate for patient.

iv. Can have history of allogeneic HSCT transplant, but must be off immunosuppression for at least 2 wks. before enrollment and w/o GVHD and/or toxicities from HSCT.

b. Diagnosed in past 5 years w/ smoldering MM at high risk of progressing to symptomatic MM.

i. Diagnosis defined as: Bone marrow infiltration with plasma cells (PCs) ≥10% and presence of a monoclonal component, Ig G ≥3 g/dl or IgA ≥2 g/dl or Bence-Jones proteinuria >1 g/dl and absence of lytic lesions on skeletal survey, absence of hypercalcemia (corrected calcium <11 mg/dl), absence of renal failure (creatinine ≤1.5 x ULN), and absence of anemia (hemoglobin >10 g/dl or not 2 g/dl below LLN).

ii. Must meet one of following:

* ≥10% PCs in bone marrow and IgG ≥3 g/dl or IgA ≥2 g/dl,
* ≥10% PCs in bone marrow and serum FLC ratio (involved : uninvolved) >100 in blood, or
* IgG ≥3 g/dl or IgA ≥2 g/dl and FLC ratio (involved: uninvolved) >100 in blood. c. MM post-treatment disease that is clinically stable and does not require treatment at least 4 weeks prior to enrollment.

  i. At least one line of treatment and achieved at least PR by IMWG ii. Stable disease or better per IMWG based on 2 subsequent assessments at least one month apart d. history of morphologically confirmed MDS i. previously received at least one treatment for MDS, including but not limited to chemotherapy or hypomethylating agent(s). Subjects may be previously untreated if they refuse treatment with or are not appropriate candidates for chemotherapy or hypomethylating agent(s) in the investigator's opinion.

ii. intermediate, high, or very high risk MDS by IPSS-r iii. No curative intent option of allogeneic HSCT or refused consideration for allogeneic HSCT iv. Could have history of allogeneic HSCT transplant and relapsed, but must be off immunosuppression for at least 2 weeks before enrollment and without GVHD and/or toxicities from HSCT.

2. Low, moderate, to high levels of OFA expression by IHC analysis of tumor specimens.

3. HLA-A*02 haplotype.

4. ECOG performance status 0 to 2.

5. 18 years or older.

6. life expectancy ≥3 months.

7. Has following laboratory parameters w/in 28 days:

* ANC ≥500/mm3
* ALC >500/mm3
* PLT ≥25,000/mm3 and may be transfused
* Hgb >8 g/dL (may have been transfused)
* Serum creatinine ≤1.5 x ULN
* Total bilirubin ≤2.0 mg/dL, unless elevated bilirubin due to Gilbert's syndrome
* ALT and AST less than 5×ULN

  8. If female of child-bearing potential, negative serum pregnancy test result w/in 28 of D1 and agree to abstain from heterosexual intercourse or use acceptable method of birth control (hormonal or barrier method) from Screening through 30 days after last dose

  9. If male having sexual contact with a female of child-bearing potential, agrees to use a latex condom dor agrees to ensure partner uses an acceptable method of birth control (hormonal or barrier method)from Screening through 30 days after last dose

  10. Able to provide written informed consent

Exclusion Criteria

1. Received chemotherapy, biological therapy, or radiation therapy less than one month before D1
2. No prior history of active CNS involvement
3. Grade 2 or higher peripheral neuropathy w/in 28 days
4. Acute promyelocytic leukemia (FAB M3)
5. Other active systemic malignancy treated w/ cytotoxic chemotherapy in previous 12 mos.
6. Monoclonal gammopathy of undetermined significance
7. For smoldering MM, baseline bone lesions or plasmacytomas
8. For smoldering MM, lytic lesions on skeletal surveys and hypercalcemia (i.e., ≥11 mg/dL)
9. Known HIV or hepatitis virus infection
10. Active infection requiring antibiotics
11. History of prior or active autoimmune disease such as Lupus or rheumatoid arthritis
12. Significant kidney or liver disease, uncontrolled severe cardiovascular or pulmonary disease, other uncontrolled medical condition that would compromise subject's ability to tolerate study treatment
13. Received any investigational treatment w/in 30 days
14. Receiving systemic glucocorticosteroid >10 mg daily. Concurrent use after registration on study should be restricted to equivalent of prednisone 10 mg per day. Prior or concurrent topical or localized glucocorticosteroid therapy to treat non-malignant comorbid disorders is permitted. Subject requiring routine use of steroid inhalers are not eligible.
15. Major surgery w/in 4 wks.
16. G-CSF w/in 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Determine the safety, dose-limiting toxicity (DLT), maximum tolerated dose (MTD), and optimal biologic dose (OBD) of BB-MPI-03 and adjuvants in subjects with hematologic cancers who are off treatment and with stable disease (SD) or better. | 6 months treatment, 6 months follow-up
  The safety and tolerability of BB-MPI-03 in Montanide emulsion preceded by sargramostim will be measured by:
  * The proportion of subjects experiencing adverse events (AEs), serious adverse events (SAEs), DLTs, and AEs leading to study vaccine discontinuation.
  * The proportion of subjects requiring a modification of the study treatment dose or schedule.
  * Change from baseline in absolute neutrophil counts (ANC) and platelet counts.
  * The proportion of subjects with local injection site reactivity.
  * Proportion of subjects experiencing infections or fevers requiring hospitalization and/or intravenous (IV) antibiotics.

SECONDARY OUTCOMES:
Determine the in vivo cellular immune response profile of BB-MPI-03 and adjuvants in subjects who receive 5 and 6 intradermal (ID) injections over a 6- month period. | 12 Months
  Immunologic responses (change from Baseline) will be assessed by:
  * DTH reaction to the peptides, as measured and photographed at 7 months using the "ballpoint pen" method.
  * Peptide-specific T-cell proliferation to ELISPOT and tetramer assay.
  * Level of OFA expression on tumor cells at Month 7.
  * Anti-peptide (anti-OFA) antibodies in the serum. These parameters will be measured at D15, D29, M2, M3, M6, M9, and M12 and compared to pre-treatment Baseline. DTH reaction to the peptides and OFA expression will be measured and recorded at 1 month after the last injection (M7).
Evaluate any anti-tumor activity of BB-MPI-03 and adjuvants as assessed by disease reduction and lack of disease progression during and after treatment. | 12 Months
  The anti-tumor activity of BB MPI 03 in Montanide emulsion preceded by sargramostim will be measured by:
  Time to progression (TTP) Overall response rate at Month 7 Best Overall Response

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Virginia Cancer Specialists, Fairfax, Virginia